CLINICAL TRIAL: NCT02815878
Title: Project Enhance for Adults Aging With Long-Term Physical Disability
Brief Title: Enhance Wellness for Individuals With Long-Term Physical Disabilities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Ivan Molton, Associate Professor, Rehabilitation Medicine, University of Washington
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 47035
Record Dates: First submitted 2016-06-22; First posted 2016-06-28 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2017-10

CONDITIONS: Multiple Sclerosis; Muscular Dystrophy; Post-polio Syndrome; Spinal Cord Injury
MeSH Terms: conditions — Multiple Sclerosis; Muscular Dystrophies; Postpoliomyelitis Syndrome; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: Intervention with Disability (Experimental): Participants with a diagnosis of multiple sclerosis, spinal cord injury, muscular dystrophy, or post-polio syndrome aged 45 or older receive Enhance Wellness for 6 months and complete pre and post outcome assessments.
  Interventions: Behavioral: Enhance Wellness
- Group 2: Intervention without Disability (Active Comparator): Participants without a diagnosis of multiple sclerosis, spinal cord injury, muscular dystrophy, or post-polio syndrome aged 45 or older receive Enhance Wellness for 6 months and complete pre and post outcome assessments.
  Interventions: Behavioral: Enhance Wellness
- Group 3: No intervention (No Intervention): Participants with a diagnosis of multiple sclerosis, spinal cord injury, muscular dystrophy, or post-polio syndrome aged 45 or older complete pre and post outcome assessments.

INTERVENTIONS:
Behavioral: Enhance Wellness — A 6-month health promotion intervention which pairs participants with a wellness coach to identify and pursue a health-related goal of their choosing.
  Arms: Group 1: Intervention with Disability; Group 2: Intervention without Disability

SUMMARY:
This project is an adaptation trial, testing the efficacy of an evidence-based community wellness program, Enhance Wellness (http://www.projectenhance.org/enhancewellness.aspx), in a sample of middle and older-aged adults living with multiple sclerosis, spinal cord injury, post-polio syndrome and muscular dystrophy.

DETAILED DESCRIPTION:
This is a quasi-experimental project, comparing the effects of Enhance Wellness in a sample of adults aged 45 years or older and living with long-term physical disability, to two quasi-control groups: a sample of adults without long-term disability participating in Enhance Wellness, and a sample of adults with long-term disability not participating in Enhance Wellness. Outcomes are collected pre-intervention and post-intervention, approximately 6-months apart.

ELIGIBILITY:
Inclusion Criteria:

* Multiple Sclerosis, Muscular Dystrophy, Post-Polio Syndrome, or Spinal Cord Injury diagnosis (Group 1 and 3)
* Living in King County, Washington (Group 1 only)
* Ability to read and understand English

Exclusion Criteria:

* Active suicidal ideation
* Requires the use of a mechanical ventilator to breathe or speak

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-05-12 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Questionnaire: Level of reported self-efficacy as measured by the University of Washington Self-Efficacy Scale Questionnaire | 6-months
  This is a self-reported measure of perceived efficacy to manage conditions or symptoms related to a person's physical disability or condition. Greater scores represent greater self-efficacy.
Questionnaire: Patient Reported Outcome Measurement Information System (PROMIS) Pain Interference Short Form | 6-months
  Self-reported measure of pain interference. Greater score indicate greater pain interference.
Questionnaire: Patient Reported Outcome Measurement Information System (PROMIS) Depression Short Form | 6-months
  Self-reported measure of depression. Greater scores indicated greater depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan R Molton, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No